CLINICAL TRIAL: NCT02947412
Title: Long Term Results After Sleeve Gastrectomy as a Primary Procedure in Obesity Surgery
Brief Title: Long Term Results After Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: Sana Klinikum Offenbach (Other)
Responsible Party: Principal Investigator, Sonja Chiappetta, MD, Dr. Sonja Chiappetta, Dr. Christine Stier, Prof. Rudolf Weiner, Sana Klinikum Offenbach
Other Study IDs: FF 1/2016
Record Dates: First submitted 2016-10-26; First posted 2016-10-27 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Obesity
Keywords: sleeve gastrectomy; long-term follow-up; gastroesophageal reflux disease after sleeve; revisional surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- sleeve gastrectomy: laparoscopic sleeve gastrectomy
  Interventions: Other: laparoscopic sleeve gastrectomy

INTERVENTIONS:
Other: laparoscopic sleeve gastrectomy — laparoscopic sleeve gastrectomy

SUMMARY:
Today sleeve gastrectomy is the most performed bariatric procedure worldwide. Since 2005 it is gaining popularity as a single procedure. Long term data is scarce. In this retrospective study long term follow-up in relation to weight loss, comorbidities, re-do and revisional surgery is getting analyzed.

DETAILED DESCRIPTION:
Today sleeve gastrectomy is the most performed bariatric procedure worldwide. Since 2005 it is gaining popularity as a single procedure. Long term data is scarce.

Re-Do and revisional surgery in form of re-sleeve, gastric bypass (mini -gastric bypass, roux-en y gastric bypass) and biliopancreatic diversion (BPD) is described in the current literature due to weight regain and reflux. The investigators want to analyze the frequency of this re-do/revisional surgery and want to compare weight loss and improvement in comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* s.a. sleeve gastrectomy since 2007

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent sleeve gastrectomy since 2007, being the first szrgical treatment for severe obesity are studied in the long term follow-up
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-01; Primary Completion 2015-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Incidence of revisional surgery | up to 9 years after surgery

SECONDARY OUTCOMES:
Excess weight loss in % | up to 9 years after surgery
Incidence of Gastroesophageal Reflux Disease | up to 9 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf A Weiner, Prof., Study Director — Sana Klinikum Offenbach

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biter LU, Gadiot RP, Grotenhuis BA, Dunkelgrun M, van Mil SR, Zengerink HJ, Smulders JF, Mannaerts GH. The Sleeve Bypass Trial: a multicentre randomized controlled trial comparing the long term outcome of laparoscopic sleeve gastrectomy and gastric bypass for morbid obesity in terms of excess BMI loss percentage and quality of life. BMC Obes. 2015 Aug 26;2:30. doi: 10.1186/s40608-015-0058-0. eCollection 2015. PMID 26316928
- [Background] Sarela AI, Dexter SP, O'Kane M, Menon A, McMahon MJ. Long-term follow-up after laparoscopic sleeve gastrectomy: 8-9-year results. Surg Obes Relat Dis. 2012 Nov-Dec;8(6):679-84. doi: 10.1016/j.soard.2011.06.020. Epub 2011 Jul 20. PMID 21890430
- [Result] Abelson JS, Afaneh C, Dolan P, Chartrand G, Dakin G, Pomp A. Laparoscopic Sleeve Gastrectomy: Co-morbidity Profiles and Intermediate-Term Outcomes. Obes Surg. 2016 Aug;26(8):1788-93. doi: 10.1007/s11695-015-2002-2. PMID 26660488
- [Result] Ramos AC, Bastos EL, Ramos MG, Bertin NT, Galvao TD, de Lucena RT, Campos JM. MEDIUM-TERM FOLLOW-UP RESULTS WITH LAPAROSCOPIC SLEEVE GASTRECTOMY. Arq Bras Cir Dig. 2015;28 Suppl 1(Suppl 1):61-4. doi: 10.1590/S0102-6720201500S100017. PMID 26537277
- [Result] Perrone F, Bianciardi E, Benavoli D, Tognoni V, Niolu C, Siracusano A, Gaspari AL, Gentileschi P. Gender Influence on Long-Term Weight Loss and Comorbidities After Laparoscopic Sleeve Gastrectomy and Roux-en-Y Gastric Bypass: a Prospective Study With a 5-Year Follow-up. Obes Surg. 2016 Feb;26(2):276-81. doi: 10.1007/s11695-015-1746-z. PMID 26033435